CLINICAL TRIAL: NCT04995718
Title: Intelligent Physical Exercise Training (IPET) in the Offshore Wind Industry: A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Ørsted A/S (Unknown)
Responsible Party: Principal Investigator, Anne Skov Oestergaard, Principal Investigator, University of Southern Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S-20182000-161
Record Dates: First submitted 2021-07-15; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-07

CONDITIONS: Physical Capacity
Keywords: Physical Capacity; Feasibility; Workplace exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IPET: Intelligent physical exercise training during working hours (Experimental): Workplace physical exercise
  Interventions: Other: Intelligent Physical Exercise Training (IPET)

INTERVENTIONS:
Other: Intelligent Physical Exercise Training (IPET) — Wind technicians performed 1-hour weekly individualized physical exercise training during working hours. The specific content of the exercise program was based on the specific job exposure profile, the physical capacity profile and the physical health profile of the employee.

SUMMARY:
A study to assess the feasibility of a 12-week exercise intervention aiming at improving the physical capacity and health of wind technicians.

it was hypothesized that the intervention would be well-accepted by workers and show high compliance and clinically relevant increases in physical capacities among wind technicians.

DETAILED DESCRIPTION:
One-arm feasibility study, including a within-group control period, to test compliance, practicality, acceptability and preliminary efficacy of implementing intelligent physical exercise training (IPET) in the offshore wind industry among wind technicians. The exercise program was individually tailored based on the findings from a pre-screening health and physical capacity check and the occupational demands of wind technicians. Primary outcomes were compliance, adherence, adverse events and satisfaction. Secondary outcomes were physical capacity and musculoskeletal disorders. Prior to the feasibility study, intervention mapping was used as a theoretical tool to plan the intervention. The intervention consisted of 1-hour weekly individually tailored exercise training during working hours. Exercise sessions were supervised during the first 8 weeks of the intervention and self-administered the last 4 weeks. The design included a 6 month control period prior to initiating the intervention. Thus, included technicians (n:24) had their health and physical capacity assessed 6 months prior to intervention start (T1), at intervention start (T2) and 12 weeks after (T3) and they responded to questionnaires on musculoskeletal symptoms at all three occasions. Further, a questionnaire customized to the specific intervention was distributed to all technicians 8 weeks after intervention start to assess satisfaction with the exercise program.

ELIGIBILITY:
Inclusion Criteria:

Wind technician Valid fitness and medical certificate Adult >18 years

Exclusion Criteria:

Hypertensive with blood pressure above 165 mmHg systolic and 105 mmHg diastolic.

Severe pain would exclude technicians from strength measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Compliance | From T2 to T3 (three months)
  The appointed supervisors tracked compliance during the first 8 weeks of the exercise intervention (192 possible sessions) on behalf of all participants. Compliance was recorded if a WT attended the planned (and facilitated) session and is reported in percentage of possible sessions.
  During the last four weeks (self-administered exercise), participants were asked to report attendance in a similar way by phone to the supervisor or health and safety representative or by filling out a record located at the onshore facility. Missing reportings were interpreted as non-compliance.
Acceptability | One time after 8 weeks (between T2 and T3)
  Acceptability with the on-site part of the intervention was evaluated after the first 8 weeks using a survey customised to the intervention and to the specific target group. Questions concerned overall acceptability and satisfaction with workplace exercise programmes in general and the specific content of this intervention. Responses were reported on a 5-point Likert scale (from "Strongly disagree" to Strongly agree")
Adherence | From T2 to T3 (three months)
  The appointed supervisors tracked adherence during the first 8 weeks of the exercise intervention (192 possible sessions) on behalf of all participants. Adherence was reached and reported if the WT completed the exercise programme as prescribed, meaning that they did not deviate from the structure of the individual exercise programme (exercise selection (or approved alternative exercises), volume and intensity). Adherence is reported in percentage of possible sessions.
  During the last four weeks (self-administered exercise), participants were asked to report attendance in a similar way by phone to the supervisor or health and safety representative or by filling out a record located at the onshore facility. Missing reportings were interpreted as non-adherence.
Adverse events | From T2 to T3 (three months)
  Supervisors were asked to record mild (e.g. soreness beyond expected levels) and serious adverse events (safety related incidents, e.g. dropped objects and sprains/strains associated with conducting the exercises) related to the training sessions. Adverse events were reported in absolute numbers.

SECONDARY OUTCOMES:
Cardiovascular capacity | Nine months (changes between T1, T2 and T3)
  Cardiovascular capacity tests were conducted at three time points: T1 (6 months prior to intervention start), T2 (intervention start) and T3 (after 12 weeks).
  Cardiovascular capacity (relative VO2max expressed in ml O2/kg/min) was indirectly assessed using the submaximal Chester Step Test on a 30 cm step.
Muscle strength | Nine months (changes between T1, T2 and T3)
  Muscle strength measurements were performed as maximal voluntary contractions of the forearm using a hand grip dynamometer and isometric shoulder abduction using hand-held dynamometry. Forearm and shoulder strength were assessed three times for the dominant arm and the maximal values were reported in kilos as means +/- SD.
Musculoskeletal disorders | Nine months (changes between T1, T2 and T3)
  Musculoskeletal disorders were assessed in terms of prevalence and severity for 9 different body parts using the Nordic Musculoskeletal Questionnaire, and cases were included if WTs had experienced symptoms for more than 1 day and with an average symptom severity of ≤ 1 (0-10) within the past 3 months.
Work ability | Nine months (changes between T1, T2 and T3)
  Singe-item from the work ability index assessing current work ability compared to lifetime best an 11-point scale (0-10). Reported as mean +/- SD
Physical fitness capacities | Nine months (changes between T1, T2 and T3)
  The validated Strøyer-scale assessing 5 items (aerobic fitness, muscle strength, endurance, flexibility and balance) on a 10 point-scales (1-10), with 1 indicating 5 indicating average physical capacity compared with peers.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Søgaard, PhD, Principal Investigator — University of Southern Denmark
Locations (1):
- Physical Activity and Health at Work, Department of Sports Science and Clinical Biomechanics, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oestergaard AS, Sandal LF, Smidt TF, Sogaard K. Intelligent Physical Exercise Training (IPET) in the offshore wind industry: a feasibility study with an adjusted conceptual model. Pilot Feasibility Stud. 2022 Jul 23;8(1):152. doi: 10.1186/s40814-022-01106-z. PMID 35870979